CLINICAL TRIAL: NCT04347174
Title: A Clinical Trial to Evaluate the Safety and Efficacy of Mycobacterium W in Critically Ill Patients Suffering From COVID 19 Infection
Brief Title: A Clinical Trial of Mycobacterium w in Critically Ill COVID 19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cadila Pharnmaceuticals (Industry)
Collaborators: Council of Scientific and Industrial Research, India (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRSC20004
Record Dates: First submitted 2020-03-31; First posted 2020-04-15 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized, blinded, two arms, active comparator controlled, clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator, patient and study staff will be blinded to the study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suspension of Mw + Standard therapy of COVID-19 (Experimental): 0.3 ml (0.1ml x 3 Injection) of intradermal Mw for 3 consecutive days
  + Standard therapy of COVID-19
  Interventions: Drug: Suspension of heat killed (autoclaved) Mycobacterium w
- Standard therapy of COVID-19 (Placebo Comparator): 0.3 ml (0.1ml x 3 Injection) of Placebo intra-dermal for 3 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suspension of heat killed (autoclaved) Mycobacterium w — Patients will be randomized to receive either Mycobacterium w in combination with standard care as per hospital practice or standard care alone in COVID-19 as per hospital practice.
  Other Names: Standard care of treatment for COVID-19 as per hospital practice
  Arms: Suspension of Mw + Standard therapy of COVID-19
Drug: Placebo — All patients will continue to receive standard therapy as per hospital practice till considered requisite by the treating physician
  Other Names: Standard care of treatment for COVID-19 as per hospital practice
  Arms: Standard therapy of COVID-19

SUMMARY:
The trial is randomized, blinded, two arms, active comparator controlled, clinical trial to evaluate the safety and efficacy of Mycobacterium w in combination with standard care as per hospital practice versus standard care alone in critically ill adult patients suffering from COVID-19 infection.

DETAILED DESCRIPTION:
In this study, Eligible patients will be enrolled after due consent and will be randomized in balance to receive either test drug (along with the standard of care) or Placebo (along with the standard of care). The enrolled patients will be monitored for any adverse events (AEs) or serious adverse events (SAEs) throughout the study period. All patients will continue to receive standard therapy till considered requisite by the treating physician.

In addition to the standard care for COVID-19, patients randomized to test arm will receive single daily dose of 0.3 ml of Mw, intradermal, for 3 consecutive days while patients randomized to control arm will receive single daily dose of 0.3 ml of Placebo, intradermal, for 3 consecutive days.

Study duration for each patient will be upto 28 days post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients infected with COVID-19 (clinical/confirmed)
* Patient aged 18 years or more of either gender
* Illness of any duration with respiratory rate ≥25 breaths/minute, and at least one of the following:

  * Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.), or or
  * SpO2 ≤94% on room air, or
  * Requiring mechanical ventilation and/or supplemental oxygen
* Female patients of childbearing potential must have a negative pregnancy test within 14 days prior to first dose of study medication.
* Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedure.

Exclusion Criteria:

* Pregnant or nursing female.
* Patients with history of allergy, hypersensitivity, or any serious reaction to study medication
* Patients with a concomitant medical condition, whose participation, in the opinion of the investigator, may create an unacceptable additional risk.
* Patient previously enrolled into this study.
* Patient participating or having participated in a clinical trial with another investigational drug within the last 28 days except for investigational drugs against cancer, leukaemia or HIV.
* Patients with a life expectancy judged to be less than five days
* ALT/AST > 5 times the upper limit of normal
* Stage 4 severe chronic kidney disease or requiring dialysis (i.e. eGFR < 30)
* Patients not likely to complete the trial as per judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
7-category ordinal scale that ranges from 1 (not hospitalized with resumption of normal activities) to 7 (death) | Change in Ordinal scale from baseline to day 3, day 7, day 14, day 21 and day 28 and day of transfer from ICU, if discharged earlier than 28 days post-randomization.
  To study the effect of Mw on recovery of organ function as assessed by Ordinal scale
Sequential Organ Failure Assessment (SOFA) scores | Change in SOFA score from baseline to day 3, day 7, day 14, day 21 and day 28 and day of transfer from ICU, if discharged earlier than 28 days post-randomization.
  To study the effect of Mw on recovery of organ function as assessed by Sequential Organ Failure Assessment (SOFA) which is based on six different scores, one for each of the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems each scored from 0 to 4 with an increasing score reflecting worsening organ dysfunction

SECONDARY OUTCOMES:
Incidence of AE / SAE or event of clinical significance | Till day 28
  Any AE / SAE or event of clinical significance observed during the study.
SARS-CoV-2 detectable in nasal or oropharyngeal (OP) sample | At days 3, 7, 14, 21, and 28
  Percent of subjects with SARS-CoV-2 detectable in nasal or oropharyngeal (OP) sample.
ICU length of stay | Till day 28
  ICU length of stay
Duration of mechanical ventilation | Till day 28
  Duration of mechanical ventilation
Duration of hospitalization | Till day 28
  Duration of hospitalization
Clinical improvement | From baseline to day 14 & Day 28
  Percentage of subjects having clinical improvement defined as two-point improvement on a seven category ordinal scale.
Time (in days) from treatment initiation to death | Till day 28
  Time (in days) from treatment initiation to death.
All-cause mortality | Till day 28
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Anil Avhad, MBBS, Study Chair — Cadila Pharmaceuticals Limited
Locations (4):
- India (4):
  - All India Institute of Medical Science, Raipur, Raipur, Chhattisgarh
  - All India Institute of Medical Sciences, Bhopal, Bhopal, Madhya Pradesh
  - Postgraduate Institute of Medical Education and Research, Chandigarh
  - All lndia Institute of Medical Science, Delhi, Delhi

IPD SHARING:
Plan to Share IPD: No